CLINICAL TRIAL: NCT03666715
Title: A Multicenter Retrospective Study to Analyse the Impact of Treatment With Paliperidone Palmitate on Clinical Outcomes and Hospital Resource Utilization in Adult Patients With Schizophrenia in Portugal
Brief Title: A Study to Analyze the Impact of Treatment With Paliperidone Palmitate on Clinical Outcomes and Hospital Resource Utilization in Adult Participants With Schizophrenia in Portugal
Acronym: PsiProsper
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag Farmaceutica Ltda. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108528; R092670SCH4063 (Other: Janssen-Cilag Farmaceutica Ltda.)
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Antipsychotic Agents; Paliperidone Palmitate; Dosage Forms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Schizophrenia: Participants diagnosed with schizophrenia who switched from oral antipsychotics (OAPs) to Paliperidone Palmitate 1-month formulation (PP1M), with available information concerning the annual schizophrenia-related hospitalizations before and after initiation of PP1M treatment, and who switched to PP1M at least 6-months after it was available for reimbursement in Portugal will be observed. The primary data source for this study will be the medical records of each participant.
  Interventions: Drug: Oral Antipsychotics (OAPs); Drug: Paliperidone Palmitate 1-Month Formulation (PP1M)

INTERVENTIONS:
Drug: Oral Antipsychotics (OAPs) — No study treatment will be administered as a part of this study. Participants will receive OAPs (such as olanzapine, risperidone, paliperidone, aripiprazole or quetiapine) as per their usual clinical practice.
Drug: Paliperidone Palmitate 1-Month Formulation (PP1M) — No study treatment will be administered as a part of this study. Participants will receive PP1M as per their usual clinical practice.

SUMMARY:
The purpose of this study is to investigate the mean number of schizophrenia-related hospital admissions, in adult participants with schizophrenia, occurred during 12 months before and 12 months after initiation of Paliperidone Palmitate 1-month formulation treatment.

ELIGIBILITY:
Inclusion Criteria:

* Must have a confirmed diagnosis schizophrenia according to the International Classification of Diseases (ICD) 9th Edition codes, or the correspondent ICD-10 codes if applicable
* Must have been treated with oral antipsychotics (OAPs) and who switched to paliperidone palmitate 1-month formulation (PP1M) due to poor adherence, or lack of efficacy (no significant symptom reduction, as judged by the treating physician, at maximum recommended dose of an antipsychotic for 6 weeks), or participants' choice, or unknown reason when the switch has not been clearly justified
* Had been treated with OAPs for at least 12 months prior to switching to PP1M. During the treatment with OAPs, dose adjustments were allowed. Participants should have been treated with PP1M for at least 4 consecutive months after the switch
* Must have available information concerning the annual schizophrenia-related hospitalizations before and after initiation of PP1M treatment during the observation period, and with the indication of PP1M initiation in their medical charts
* Must be being treated at an ambulatory setting at study entry

Exclusion Criteria:

* Participants with schizophrenia resistant to treatment (TR). TR is defined for the purpose of this study by at least two failed adequate trials with different antipsychotics (at maximal antipsychotic efficacious label dose for 4 to 6 consecutive weeks)
* Participants that used clozapine as treatment for schizophrenia in any given period prior to or during the observation period, independently of other concomitant psychotropic medication
* Participants who have participated in a clinical trial during the observation period
* Participants that switched to PP1M before the 31st of July 2014, that is in the first 6 months after it was available for reimbursement in Portugal

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population will include ambulatory participants diagnosed with schizophrenia that switched from oral antipsychotics (OAPs) to paliperidone palmitate 1-month formulation (PP1M), and with available information concerning the annual schizophrenia-related hospitalizations before and after initiation of PP1M treatment.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Mean Number of Schizophrenia-Related Hospital Admissions Occurred During 12 Months of OAP Treatment Prior to PP1M Treatment | Approximately 12 months
  Mean number of schizophrenia-related hospital admissions occurred during 12 months of oral antipsychotics (OAP) treatment prior to initiation of Paliperidone Palmitate 1-Month Formulation (PP1M) treatment will be reported. Mean number of Schizophrenia-related hospital admissions will be calculated as: number of hospital admissions divided by total number of participants.
Mean Number of Schizophrenia-Related Hospital Admissions Occurred During 12 Months After Initiation of PP1M Treatment | Approximately 12 months
  Mean number of schizophrenia-related hospital admissions occurred during 12 months after initiation of PP1M treatment will be reported. Mean number of Schizophrenia-related hospital admissions will be calculated as: number of hospital admissions divided by total number of participants.
Mean Change of Schizophrenia-Related Hospital Admissions Between Periods | Approximately 24 months
  Mean change of schizophrenia-related hospital admissions occurred between periods (during 12 months of OAP treatment prior and 12 months after initiation of PP1M treatment) will be reported.

SECONDARY OUTCOMES:
Mean Number of Hospital Admissions Occurred During 12 Months of OAP Treatment Prior to PP1M and During 12 Months After Initiation of PP1M Treatment for the Subgroup of Participants that Completed 12 Months of PP1M Treatment | Approximately 24 months
  Mean number of hospital admissions occurred during 12 months of OAP treatment prior to PP1M and during 12 months after initiation of PP1M treatment for the subgroup of participants that completed 12 months of PP1M treatment will be reported. Mean number of hospital admissions will be calculated as: number of hospital admissions divided by total number of participants.
Mean Change of Hospital Admissions Between Periods for the Subgroup of Participants that Completed 12 Months of PP1M Treatment | Approximately 24 months
  Mean change of hospital admissions occurred for the subgroup of participants that completed 12 months of PP1M between periods (during 12 months of OAP treatment prior and after initiation of PP1M treatment) will be reported.
Mean Number of Hospital Admissions Occurred During 12 Months of OAP Treatment Prior to PP1M and During 12 Months After Initiation of PP1M Treatment for the Subgroup of Participants that Discontinued Before Completing 12 Months of PP1M Treatment | Approximately 24 months
  Mean number of hospital admissions occurred during 12 months of OAP treatment prior to PP1M and during 12 months after initiation of PP1M treatment for the subgroup of participants that discontinued before completing 12 months of PP1M treatment will be reported. Mean number of hospital admissions will be calculated as: number of hospital admissions divided by total number of participants.
Mean Change of Hospital Admissions Between Periods for the Subgroup of Participants That Discontinued Before Completing 12 Months of PP1M Treatment | Approximately 24 months
  Mean change of hospital admissions occurred for the subgroup of participants that discontinued before completing 12 months of PP1M treatment between periods (during 12 months of OAP treatment prior and after initiation of PP1M treatment) will be reported.
Mean Length of Hospitalizations | Approximately 24 months
  Mean length of hospitalizations occurred during 12 months after initiation of OAP treatment and the mean length of hospitalizations occurred during 12 months after initiation of PP1M treatment will be reported.
Mean Change in Length of Hospitalizations Between Periods | Approximately 24 months
  Mean change in length of hospitalizations between periods (occurred during 12 months after initiation of OAP treatment and during 12 months after initiation of PP1M treatment) will be reported.
Mean Cumulative Length of Hospitalizations | Approximately 24 months
  The mean cumulative length of hospitalizations occurred during 12 months after initiation of OAP treatment and the mean length of hospitalizations occurred during 12 months after initiation of PP1M treatment will be reported.
Mean Change in Cumulative Length of Hospitalizations Between Periods | Approximately 24 months
  Mean change in cumulative length of hospitalizations between periods (occurred during 12 months after initiation of OAP treatment and during 12 months after initiation of PP1M treatment) will be reported.
Hospitalization Rate per Patient-Years | Approximately 24 months
  The hospitalization rate per patient-year will be calculated as: Hospitalization rate per patient-years = Number of hospitalizations in the treatment period divided by total follow-up time in the treatment period where the total follow-up time corresponds to the cumulative follow-up time of all included participants in the treatment period.
Mean Number of Emergency Psychiatric Visits | Approximately 24 months
  The mean number of emergency psychiatric visits occurred during 12 months of OAP treatment prior to PP1M and the mean number of emergency psychiatric visits occurred during 12 months after initiation of PP1M treatment will be reported.
Mean Change in Emergency Psychiatric Visits Between Periods | Approximately 24 months
  Mean change in emergency psychiatric visits between periods (occurred during 12 months of OAP treatment prior to PP1M and during 12 months after initiation of PP1M treatment) will be reported.
Percentage of Participants Hospitalized | Approximately 24 months
  Percentage of participants hospitalized during 12 months of OAP treatment prior to PP1M and the percentage of participants hospitalized during 12 months after initiation of PP1M treatment will be reported.
Change in Percentages of Participants Hospitalized Between Periods (Hospitalization Reduction Percentage) | Approximately 24 months
  Change in percentage of participants hospitalized between periods (percentage of participants hospitalized during 12 months of OAP treatment prior to PP1M and the percentage of participants hospitalized during 12 months after initiation of PP1M treatment) will be reported.
Percentage of Outpatient Psychiatric Consultations | Approximately 24 months
  Percentage of outpatient psychiatric consultations occurred during 12 months of OAP treatment prior to PP1M and the percentage of outpatient psychiatric consultations occurred during 12 months after initiation of PP1M treatment will be reported.
Change in Percentage of Outpatient Psychiatric Consultations Between Periods | Approximately 24 months
  Change in percentage of outpatient psychiatric consultations between periods (occurred during 12 months of OAP treatment prior to PP1M and during 12 months after initiation of PP1M treatment) will be reported.
Percentage of Relapse with Different Causes | Approximately 24 months
  Percentage of relapse with different causes occurred during 12 months of OAP treatment prior to PP1M and the percentage of relapse occurred during 12 months after initiation of PP1M treatment will be reported.
Change in Percentages of Relapse Between Periods with Different Causes | Approximately 24 months
  Change in percentage of relapse between periods with different causes (occurred during 12 months of OAP treatment prior to PP1M and during 12 months after initiation of PP1M treatment) will be reported.
Percentage of Participants who Discontinued PP1M Treatment with Different Reasons for Discontinuation Before and After Completing 12 Months of Treatment | Approximately 24 months
  Percentage of participants who discontinued PP1M treatment with different reasons for discontinuation (such as, lack of efficacy, tolerability issues or other) before and after completing 12 months of treatment will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Farmaceutica Ltda. Clinical Trial, Study Director — Janssen-Cilag Farmaceutica Ltda.
Locations (1):
- Neurobios , Instituto De Neurociências, Porto, Portugal